CLINICAL TRIAL: NCT07270601
Title: Development and Diagnostic Evaluation of a Novel Quantifiable Ultrasound Based Multi-parametric Biomarker for Hepatic Steatosis in Patients With Suspected MASLD ( LYNX )
Brief Title: Development of a Quantifiable Ultrasound Biomarker for Hepatic Steatosis
Acronym: LYNX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ContextVision AB (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COV-POCUS-001
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; NAFLD - Non-Alcoholic Fatty Liver Disease
Keywords: MASLD; NAFLD; Ultrasound; Steatosis; Fibrosis; MRI-PDFF
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cohort (Experimental): Adult healthy volunteers as well as subjects who have a diagnosis, or suspected, of having MASLD or are deemed to meet the high-risk cardiometabolic criteria.
  Interventions: Device: Verasonics NXT Data Acquisition System; Device: Philips EPIQ Elite; Device: EchoSense FibroScan; Device: Philips 3T Ingenia Elition

INTERVENTIONS:
Device: Verasonics NXT Data Acquisition System — A research ultrasound imaging device to capture raw radiofrequency ultrasound data for the following parameters:
  * B-mode imaging
  * Attenuation coefficient
  * Backscatter coefficient
  * Speed of sound
  * Shear wave elastography
Device: Philips EPIQ Elite — A premium ultrasound system with software package to support imaging research studies.
Device: EchoSense FibroScan — A non-invasive ultrasound solution that accurately measures liver stiffness and liver steatosis.
Device: Philips 3T Ingenia Elition — A 3-tesla magnetic resonance imaging (MRI) system

SUMMARY:
The research study is considering a non-invasive way to measure the percentage of fat in the liver using ultrasound. This could help detect early signs of a very common condition called metabolic dysfunction-associated steatotic liver disease (MASLD). Current tests, like MRI or biopsy, can be expensive or invasive. If successful, this ultrasound tool could become an easier and more accessible way to monitor liver health - especially for people with obesity, diabetes, high blood pressure, or high cholesterol.

DETAILED DESCRIPTION:
The objective is to develop a novel multiparametric ultrasound-based technique to quantify the amount of steatosis in the liver by using the current MRI-based gold-standard - MRI proton density fat fraction (MRI-PDFF) as a clinical reference. This clinical development study will only collect the required dataset from healthy volunteers and subjects with different degrees of steatosis in the liver, particularly patients with MASLD, formerly non-alcoholic fatty liver disease (NAFLD). It will capture the raw radiofrequency data required for the development of this new radiologic biomarker on a research ultrasound imaging device. In addition, various other clinical and radiological datasets will be captured to support the ground truthing, development and training of the novel ultrasound-based multiparametric biomarker.

ELIGIBILITY:
Inclusion Criteria:

Diseased subject:

* Adult patients (age 18 - 75 years)
* Consent to participate in the study
* Diagnosed or suspected MASLD from the hepatology clinic, OR
* High-risk population meeting the adult cardiometabolic criteria (defined as the presence of at least one of the following: diabetes, obesity (BMI ≥ 25 kg/m2), hypercholesterolemia, and hypertension)

Healthy volunteer:

* Adult patients (age 18 - 75 years)
* Consent to participate in the study
* No suspicion of MASLD by laboratory/imaging/clinical examinations
* Absence of known pre-existing conditions (metabolic syndrome, diabetes mellitus, obesity, insulin resistance, dyslipidemia, etc.)

Exclusion Criteria:

* Pregnancy or nursing.
* Contraindications to MRI including, but not limited to, severe claustrophobia, pacemaker, or existing metallic/mechanical implant(s).
* Acute illness/cognitive impairment resulting in an inability to cooperate with the MRI and ultrasound breath-holding instructions.
* BMI > 35 kg/m2
* History of excessive alcohol consumption according to the updated MASLD criteria (>2 drinks/day OR >210 grams/week for males AND >1 drink/day OR >140 grams/week for females) or drug use over the past 2 years.
* Known acute or chronic hepatitis; or other etiology of liver disease.
* Presence of known congenital hepatic anomaly.
* Known cirrhosis
* Known active cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Multiparametric Ultrasound Biomarker vs. MR-PDFF | 1 year
  Clinical qualification of the multiparametric ultrasound-derived fat fraction, defined as its agreement with the established clinical reference, MRI proton density fat fraction (MRI-PDFF) expressed as absolute percentage, in bench testing analysis.

SECONDARY OUTCOMES:
Individual Ultrasound parameter vs. MRI-PDFF | 1 year
  Evaluation of each ultrasound parameter (backscatter, attenuation and speed of sound) fat percentage values separately against MRI-PDFF.
Ultrasound Shear Wave vs MR Elastography | 1 year
  Evaluation of ultrasound shear wave elastography-derived tissue stiffness values in kilopascals compared to MR elastography.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No